CLINICAL TRIAL: NCT07186933
Title: Driving Pressure During Surgeries With High Risk for Postoperative Pulmonary Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University General Hospital of Patras (Other)
Responsible Party: Principal Investigator, Antonios Kostouros, Prinsipal Investigator, Antonios Kostouros, University General Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22624 / 4.8.2025
Record Dates: First submitted 2025-08-20; First posted 2025-09-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pulmonary Atelectasis; Postoperative Pulmonary Complications; Postoperative Respiratory Failure; Postoperative Bronchospasm; Postoperative Pleural Effusion; Postoperative Pneumothorax; Postoperative Pneumonia; Postoperative Aspiration Pneumonitis; Mechanical Power; Driving Pressure
Keywords: Driving Pressure; Mechanical Power; Atelectasis; Pulmonary Complications; Postoperative Pulmonary Complications; Postoperative Respiratory Failure; Elastic Power
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Protective Ventilation (Other): CONVENTIONAL LUNG PROTECTIVE VENTILATION
  This group is mechanically ventilated with Invasive Mechanical Ventilation with PEEP 8 cm H20 Tidal Volume (VT) 8 ml/kg Ideal Body Weight (IBW) Respiratory Rate (RR) --> Arterial Partial CO2 Pressure (PaCO2) = 35-45 mmHg Inspired Oxygen Fracture (FiO2) 0.4 - 0.5 --> Peripheral Oxygen Saturation (SpO2) > 93% Recruitment Maneuver (as described) every hour
  Interventions: Procedure: Lung Protective Ventilation
- Minimum Driving Pressure (Active Comparator): This group is mechanically ventilated with Invasive Mechanical Ventilation with PEEP; Initially 8 cm H2. Titrated at level with Minimum Driving Pressure after first recruitment - titration maneuver followed by new recruitment maneuver VT 8 ml/kg IBW RR --> PaCO2 = 35-45 mmHg FiO2 0.4 - 0.5 --> SpO2 > 93% Recruitment Maneuver (as described) every hour
  Interventions: Procedure: PEEP titration for Minimum Driving Pressure

INTERVENTIONS:
Procedure: PEEP titration for Minimum Driving Pressure — This group is mechanically ventilated with Invasive Mechanical Ventilation with Volume Control Ventilation mode with PEEP Initially 8 cm H2O. Afterwards, the lungs are recruited with the aforementioned maneuver. During subsequent derecruitment, PEEP is decreased by 2 cm H20 and compliance is noted in each stage. The goal is to find PEEP with maximum compliance (Cmax). A new recruitment maneuver follows and during derecruitment PEEP is set at the optimum value that was previously defined.
  VT 8 ml/kg IBW RR --> PaCO2 = 35-45 mmHg FiO2 0.4 - 0.5 --> SpO2 > 93% Recruitment Maneuver (as described) every hour
  Other Names: Maximum compliance mechanical ventilation; Cmax Mechanical Ventilation
  Arms: Minimum Driving Pressure
Procedure: Lung Protective Ventilation — This group is mechanically ventilated with Invasive Mechanical Ventilation with Volume Control Ventilation mode with PEEP 8 cm H2O. VT 8 ml/kg IBW RR --> PaCO2 = 35-45 mmHg FiO2 0.4 - 0.5 --> SpO2 > 93% Recruitment Maneuvers (as described) every hour
  Arms: Lung Protective Ventilation

SUMMARY:
The goal of this clinical trial is to compare two different types of perioperative mechanical ventilation (MV), specifically Protective Mechanical Ventilation (PMV) and MV with the lowest possible Driving Pressure (ΔP), in relation to the appearance of postoperative pulmonary complications (PPCs) in adult patients who are operated and have higher risk of PPCs.

The main questions it aims to answer are:

* Is MV with lower ΔP better than conventional PMV in preventing PPCs in patients with higher risk for PPCs?
* Does MV with lower ΔP decrease hospital stay, Intensive Care Unit (ICU) need and mortality?
* Does MV with lower ΔP suit better than PMV to lung characteristics and needs intraoperatively?

Researchers will compare MV with the lowest possible Driving Pressure (ΔP) to Protective Mechanical Ventilation (PMV) to see if any of this is more protective than the other concerning PPCs.

All participants will receive perioperative MV.

Half of them will receive conventional Protective Mechanical Ventilation (PMV). This will include well known generally protective settings for mechanical ventilation of patients, concerning volumes, pressures, respiratory rate, inspiratory gases and ventilation maneuvers.

The rest of participants will be ventilated with the lowest possible Driving Pressure (ΔP). This will be similar to PMV in the chosen volumes, respiratory rate, inspiratory gases and ventilation maneuvers. However, the pressure inside lung at the end of expiration, eg Positive End Expiratory Pressure (PEEP), will be not be preset for every patient. Initially, the investigators will perform a maneuver that will quantify each individual's lung characteristics and mechanics. According to this, the investigators will find the exact PEEP that seems to suit each patients lungs most, and use this perioperatively, trying to provide lungs the best conditions every time.

After the completion of the operation, all the patients will be screened for PPCs, via arterial blood testing and chest X ray, and the results will be statistically analyzed trying to find if any of the forementioned strategies of mechanical ventilation surpasses the other concerning PPCs appearance. PPCs include atelectasis, respiratory failure, bronchospasm, pleural effusion, pneumonia, aspiration and pneumothorax.

Furthermore hospital stay, ICU need and mortality will be noted. Finally, measurements of perioperative lung pressures, volumes and derived variables will be noted and compared statistically as well.

ELIGIBILITY:
Inclusion Criteria

* >17 years old
* Surgery with general anesthesia & invasive mechanical ventilation
* Preoperative ARISCAT score estimation >25

Exclusion Criteria:

* <18 years old
* Preoperative ARISCAT score estimation <26
* Women during pregnancy or just given birth
* Other type of anesthesia (Not general)
* Contraindication of administration of neuromuscular blockade agents.
* Contraindication of cease of spontaneous ventilation.
* Mechanical ventilation without endotracheal intubation.
* Severe heart failure / Severe cardiac arrhythmia.
* Severe emphysematous lung disease.
* Patient denial of participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pulmonary Complications | Atelectasis -> Within 1 hour in PACURespiratory failure -> Immediately postoperatively & after 30 minutes in PACU.Bronchospasm, Pleural Effusion, Pneumonia, Aspiration Pneumonitis, Pneumothorax -> from immediately postoperative until end of study
  Number of the following Postoperative Pulmonary Complications
  1. Postoperative Atelectasis (based on Chest X-Ray in Post-Anesthesia Care Unit - PACU)
  2. Postoperative Respiratory Failure based on Arterial Blood Gases in PACU (type I and/or II)
  3. Postoperative Bronchospasm
  4. Postoperative Pleural Effusion
  5. Postoperative Pneumonia
  6. Postoperative Aspiration Pneumonitis
  7. Postoperative Postoperative Pneumothorax

SECONDARY OUTCOMES:
Hospital Stay | From day of operation until the end of patient stay inside hospital, because of return to home or due to death.
  Total hospital stay days from day of operation until hospital discharge.
ICU need. | From day of operation until the end of patient stay inside hospital, because of return to home or due to death.
  Potential Need for ICU admission.
ICU stay | From day of operation until the end of patient stay inside hospital, because of return to home or due to death.
  In case of ICU need, total days of ICU stay.
28 Day mortality | From day of operation until up to 28 days.
  Incidence of death in 28 days in each group.
Mechanical Power (MP) | From the moment of beginning of operation until the moment of the end of operation and mechanical ventilation
  To calculate MP, the following must be recorded: RR, Peak Airway Pressure (Ppeak), Plateau Pressure (Pplat), and PEEP. The simplified equation will be used; MP = 0.098 × RR × [Ppeak - (Plat-PEEP)/2]
Volume-normalized Mechanical Power (MPcrs) | From the moment of beginning of operation until the moment of the end of operation and mechanical ventilation
  MPcrs = MP/Respiratory System Compliance (Crs)
Elastic Power (EP) | From the moment of beginning of operation until the moment of the end of operation and mechanical ventilation
  To calculate EP, the following must be recorded: RR, VT, Pplat, and PEEP. The following equation will be used: EP = 0.098 × RR × VT × [(Plat+PEEP)/2]
Volume-normalized Elastic Power (EPcrs) | From the moment of beginning of operation until the moment of the end of operation and mechanical ventilation
  EPcrs = EP/Crs

CONTACTS AND LOCATIONS:
Overall Officials: Diamanto Aretha, A. Professor, Study Director — University of Patras; Antonios Kostouros, Resident, Principal Investigator — University of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: Yes
Excel file per patient containing all the collected data Preoperatively; Patient demographics, ARISCAT score Perioperatively; Mechanical ventilation settings and measurements. Type and duration of operation. Anesthetic methods. Aerial blood gases results. Data from haemodynamic monitoring. Quantity of crystalloids , vasoperessors and inotropes.
  Postoperatively; Arterial blood gases results in PACU, Potential presence of other postoperative pulmonary complications.
  Statistic analysis of the collected data
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning at the end of data collection, possibly August 2027. Ending 3 years after publication of results.
Access Criteria: Reviewers. Researchers of relevant subjects. Anesthesiologists with interest in optimum mechanical ventilation.
  A request via email will be initially needed. A data sharing agreement will be needed to be signed.